CLINICAL TRIAL: NCT05885295
Title: Understanding Factors Affecting Cognitive Function in Cerebrovascular Disease
Brief Title: The Imperial Comprehensive Cognitive Assessment in Cerebrovascular Disease (IC3)
Acronym: IC3
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: RGIT / R&D REF: 21HH7075; MRC (Other Grant/Funding Number: P79100); 299333 (Other: IRAS); CPMS 50479 (Registry Identifier: UK CRN)
Record Dates: First submitted 2023-05-15; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Stroke (CVA) or TIA; Dementia, Vascular; Cerebrovascular Disorders; Small Vessel Cerebrovascular Disease; Cognitive Impairment
Keywords: dementia; MRI; blood biomarkers; neurofilament light; amyloid; tau; GFAP; white matter hyper intensity; micro bleed; small vessel disease; cognitive impairment; vascular dementia; stroke; aphasia; neglect
MeSH Terms: conditions — Stroke; Dementia, Vascular; Cerebrovascular Disorders; Cerebral Small Vessel Diseases; Cognitive Dysfunction; Dementia; Charcot-Marie-Tooth disease, Type 1F; Alzheimer Disease; Pick Disease of the Brain; Aphasia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patient with stroke
  Interventions: Diagnostic Test: MRI brain, Blood tests, cognitive assessments
- Controls: Age-matched controls
  Interventions: Diagnostic Test: MRI brain, Blood tests, cognitive assessments

INTERVENTIONS:
Diagnostic Test: MRI brain, Blood tests, cognitive assessments — observational study examining cognition post stroke using behavioural tests, MRI brain and blood tests

SUMMARY:
Stroke is a major cause of death and disability worldwide, frequently resulting in persistent cognitive deficits among survivors. These deficits negatively impact recovery and therapy engagement, and their treatment is consistently rated as high priority by stakeholders and clinicians. Although clinical guidelines endorse cognitive screening for post-stroke management, there is currently no gold standard approach for identifying cognitive deficits after stroke, and clinical stroke services lack the capacity for long-term cognitive monitoring and care. Currently available assessment tools are either not stroke-specific, not in-depth or lack scalability, leading to heterogeneity in patient assessments. To address these challenges, a cost-effective, scalable, and comprehensive screening tool is needed to provide a stroke-specific assessment of cognition. The current study presents such a novel digital tool, the Imperial Comprehensive Cognitive Assessment in Cerebrovascular Disease (IC3), designed to detect both domain-general and domain-specific cognitive deficits in patients after stroke with minimal input from a health professional. To ensure its reliability, we will utilise multiple validation approaches, and aim to recruit a large normative sample of age-, gender-, and education-matched UK-based controls. Moreover, the IC3 assessment will be integrated within a larger prospective observational longitudinal clinical trial, where post-stroke cognition will be examined in tandem with brain imaging and blood biomarkers to identify novel multimodal biomarkers of recovery after stroke. By leveraging this rich dataset, our study will allow more precise targeting of cognitive rehabilitation to stroke survivors that are most at risk of progressive cognitive decline and have the greatest potential for recovery.

DETAILED DESCRIPTION:
Aims and objectives

1. Develop an adaptive, scalable, self-administered, digital comprehensive cognitive screening tool to detect cognitive impairments in patients with cerebrovascular disease. The IC3 will:

   I. Detect both domain-general (e.g. executive function) and domain-specific (e.g. aphasia, apraxia, neglect) deficits post-stroke.

   II. Allow monitoring to occur at scale, in a cost-efficient manner, as test administration can occur independent of trained professionals.

   III. Minimise the effects of neglect or aphasia on cognitive assessments. IV. Have high test-re-test reliability for repeated-testing longitudinally.
2. Validate the IC3 against commonly used cognitive screening tools.
3. Apply the IC3 in a cohort of stroke survivors, as part of the main study, to map their trajectory of cognitive impairment over the course of the first year after stroke.
4. Identify novel biomarkers of cognitive outcome (cognitive scores at 1 year) and recovery trajectory through the main study using:

I. Premorbid demographics, and comorbid physical, neuropsychological and socioeconomic factors II. Structural and functional MRI brain imaging, to assess metrics of cerebrovascular disease load, stroke lesion topology and brain network dynamics.

III. Blood biomarkers of neurodegeneration (total microtubule-associated protein TAU; Phosphorylated TAU isoforms; Amyloid Aβ42/40 ratio) and neuroaxonal injury (Neurofilament Light - NFL; Glial Fibrillary Acidic protein - GFAP). The study will characterise the time course of the blood biomarkers over the first year after acute stroke and relate these to MRI measures of axonal injury and brain atrophy, as well as cognitive and functional outcomes at 12 months.

IC3 Assessment Design and Development

Cognitive tests. The IC3 assessment covers 22 short tasks, spanning a wide range of cognitive domains followed by several clinically-validated questionnaires, designed to be completed in under 60-70 minutes. IC3 is available via a web-browser on any modern device (smartphone, tablet, computer/laptop). To launch the assessment, the participant clicks on a link created by the study team.

The digital nature of the IC3 affords scalability in cognitive monitoring by being usable in both the clinical setting and home environment in the absence of a trained clinician. As well as reducing healthcare costs, this feature promotes accessibility of the assessment for physically disabled patients in whom attendance to healthcare or research setting is difficult. Compared to pen and paper tests, the IC3 test administration is standardised, scoring is automated and more detailed response metrics per individual tests are collected (e.g. capturing reaction time and trial-by-trial variability in responses, as well as accuracy). This allows real-time evaluation of cognitive impairments against normative samples of age-, education- and sex- matched controls.

Demographic and neuropsychiatric questionnaires. A number of health questionnaires and modified versions of relevant clinically-validated questionnaires are completed by the patient or carers to assess mood, apathy, fatigue and sleep.

At the end of the assessment the participant will be given a graphical, easy-to-understand diagram that highlights their performance against normative data. The normative data will be based on single time-point data collected remotely from large sample of healthy controls (>3000).

Main IC3 study design

This prospective observational longitudinal study aims to recruit 300 patients with acute stroke and obtain repeated measures of cognition and psychosocial status at baseline, 3-months, 6-months and 12-months post ictus. IC3 is currently a single-site study at Imperial College Healthcare NHS Trust, England, and commenced recruitment in 2022. In addition to the cognitive monitoring, all patients will be invited to take part in MRI brain imaging and blood biomarker sub-studies.

IC3 validation sub-study. A minimum of 100 patients will undergo clinically validated pen and paper cognitive screens. Test-retest reliability analyses will estimate the impact of learning effects on performance, and compare remote administration with in-person delivery of the assessment.

MRI sub-study. Clinically acquired brain imaging at the time of the acute stroke (including FLAIR and DWI sequences) will be obtained. All 300 patients will be invited to undergo additional brain MRI imaging at 3 and 12 months using a Siemens Verio 3T scanner at the Imperial College Clinical Imaging Facility. MRI measures will be used as prognostic indicators for cognitive trajectory.

Blood biomarkers sub-study. Blood samples will be obtained at baseline, and at 3, 6 and 12 months from 200 patients. Two EDTA (plasma) and two SST (serum) samples will be collected. Sample processing involves centrifugation at 2000g for 10 minutes at 4°C, followed by secure storage at -80°C. Additional single PAXgene sample will be collected at one time point for DNA storage for future analysis. The primary plasma biomarker of interest will be NFL. Additional markers including GFAP, total TAU, phosphorylated TAU and Amyloid Aβ42/40 ratio will be quantified. Testing will be performed at University College London via a digital ELISA technique, using a Quanterix Simoa analyser to provide ultrasensitive assessment of concentrations.

Study Population

Participant identification, recruitment and consent. Patients will be recruited from the Imperial College Healthcare NHS Trust by study personnel and the clinical team. Our goal is to recruit patients as early after stroke as is practical, and ideally within ten days to facilitate acute blood biomarker assessment. Those satisfying the inclusion and exclusion criteria will be approached and consented. If a patient is unable to provide fully informed consent, for example due to severe aphasia, we will assent with permission from a consultee. Patients that have been assented will be reconsented if they are subsequently able to provide full informed consent. The consent procedure will be carried out in strict compliance with national legislation and General Data Protection Regulation. Control participants will be aged > 18 and without history of neurological illness or serious psychiatric illness.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18
* Evidence of confirmed stroke (for patients)
* Ability to concentrate for 15 minutes at a time to engage with cognitive testing

Exclusion Criteria for the main study:

* Pre-stroke diagnosis of dementia
* Severe visuo-spatial problems, fatigue, or mental health problems
* Severe hearing impairment in the presence of reading comprehension impairment

Exclusion Criteria for the MRI imaging sub-study:

* Pregnancy
* Presence of metal implants
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with stroke
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
cognition | 1 year after stroke
  IC3-derived accuracy measures on cognitive testing Scale title: The Imperial Comprehensive Cognitive Assessment in Cerebrovascular Disease Impairment value defined as <1.5 Standard Deviation Units below the age and education -matched control sample Lower values mean worse outcome

SECONDARY OUTCOMES:
MOCA | 1 year post stroke
  Clinically derived MOCA scores for cognition Scale title: The Montreal Cognitive Assessment Range 0-30. Lower values mean worse outcome.
NIHSS | 1 year post stroke
  NIH Stroke Scale Scale title: National Institute of Health Stroke Scale Range: 0-24 Lower values mean better outcome.
Lawton and Brody Instrumental activities of daily living (IADL) | 1 year post stroke
  Scale title: Lawton and Brody Instrumental Activities of Daily Living Source: Lawton, M.P., and Brody, E.M. "Assessment living." Gerontologist 9:179-186, (1969).
  Range: 0-8 Lower values mean worse outcome.
MRS | 1 year post stroke
  Scale title: Modified Rankin Scale Range: 0-6 Lower values mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data used in publications may be shared on reasonable request from PI.

REFERENCES:
- [Derived] Gruia DC, Trender W, Hellyer P, Banerjee S, Kwan J, Zetterberg H, Hampshire A, Geranmayeh F. IC3 protocol: a longitudinal observational study of cognition after stroke using novel digital health technology. BMJ Open. 2023 Nov 24;13(11):e076653. doi: 10.1136/bmjopen-2023-076653. PMID 38000822